CLINICAL TRIAL: NCT02313402
Title: A Pilot Study Assessing a New Eye-writing Device Allowing Cursive Writing With Smooth Pursuit Eye Movements in Subjects With ALS
Brief Title: A New Eye-based Communication Device for ALS Patients
Acronym: ELY-SLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: P131101
Record Dates: First submitted 2014-12-05; First posted 2014-12-10 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-07

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EOL (Eye On Line) (Experimental): training program allowing a gradual acquisition of the eye-writing
  Interventions: Device: EOL (Eye On Line)

INTERVENTIONS:
Device: EOL (Eye On Line) — the intervention consists in training program allowing a gradual acquisition of the eye-writing

SUMMARY:
Eighteen ALS patients will be trained to control a new communication device (Eye On Line: EOL) that permit over smooth eye movements to generate digits, letters, words or drawing at will. The intervention consists in a training program during six visits over 3 weeks on site allowing a gradual acquisition of the eye-writing. The primary objective of the study is to assess the feasibility of the use of EOL device in ALS patients. The EOL device potentially offers a creative and personal means of linguistic and emotional expression in subject with motor disability.

DETAILED DESCRIPTION:
Background: Motor weakness progression in ALS challenges communication modalities such as writing or speech with a marked impairment of quality of life. In recent years the development of appropriate communication tools played a key role to maintain patients in an efficient interaction with environment and caregivers. However there is a need for tools to customize communication and provide a creative space. Eye on-line (EOL) is a new communication device with which the user is presented with an illusion inducing visual stimulus resulting in the perception of illusory movement that can be followed by the eye, so that smooth pursuit eye movement can be sustained in arbitrary directions.(1) After an appropriate training participants gain volitional control over smooth eye movements and can generate digits, letters, words or drawing at will.

Objectives: The primary objective of the study is to assess the feasibility of the use of EOL device in ALS patients. The secondary objective is to assess its clinical safety in subjects with ALS. We added exploratory objectives to evaluate eye movements in ALS patients, to study factors (neuropsychology, eye movements) that may influence the use of the apparatus and to evaluate a Bayesian computational model for online character recognition.(2) Methods: Eighteen subjects with ALS and motor impairment impairing normal writing will be recruited with a duration of participation of four weeks per patient. The intervention will consist in a training program to the device during six visits on site allowing a gradual acquisition of the ability to perform an eye-writing. The primary endpoint is the recognition by an outside observer of the digits 0-9 produced by the patient with the device. The secondary criteria is the record of adverse events and serious adverse events occurred during the study other than those directly related to ALS.

Discussion/Conclusions: EOL device potentially offers a creative and personal means of linguistic and emotional expression in subject with motor disability. The study is open to patients recruitment since June 2014. Results are expected in mid 2015.

ELIGIBILITY:
Inclusion criteria :

* 18 to 65 years old
* patient with SLA diagnosis
* patient presenting writing troubles
* patient with understandable speaking communication
* patient with health insurance

Exclusion criteria :

* patients presenting oculomotricity troubles
* patients presenting frontotemporal dementia
* patients presenting a chronic incapacitating disease other than ALS
* patients presenting epilepsy antecedents
* patents included in an other clinical study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
recognition by an outside observer of the digits 0-9 produced by the patient with the device | 4 weeks

SECONDARY OUTCOMES:
adverse events | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lucette Lacomblez, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe Hospitalier Pitie Salpetriere, Paris, France